CLINICAL TRIAL: NCT06209437
Title: The Effect of Total Intravenous Anesthesia or Inhalation Anesthesia on Inflammatory Biomarkers in Coronary Artery Bypass Surgery and Their Relationship With Early Postoperative Complications a Prospective Observational Study
Brief Title: Anesthesia Management of Coronary Artery Bypass Surgery and Inflammatory Biomarkers
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: volgaozkan1
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease; Postoperative Complications; Anesthesia
MeSH Terms: conditions — Coronary Artery Disease; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhalation Anesthesia Group: After induction, anesthesia will be provided with sevoflurane (2.0 mac) and intravenous remifentanil infusion (0.05-0.2 mcg/kg/min). Depth of anesthesia will be evaluated with Bispectral Index (BIS).
- Total Intravenous Anesthesia Group: After induction, anesthesia will be provided with intravenous propofol infusion (50-150 mcg/kg/min) and intravenous remifentanil infusion (0.05-0.2 mcg/kg/min). Depth of anesthesia will be evaluated with Bispectral Index (BIS).

SUMMARY:
The goal of this observational study is to evaluate effect of total intravenous anesthesia or inhalation anesthesia on inflammatory biomarkers in coronary artery bypass surgery and their relationship with early postoperative complications. The main questions it aims to answer are

* Does the type of anesthesia have a relationship with inflammatory biomarkers?
* Are inflammatory biomarkers associated with postoperative complications?

DETAILED DESCRIPTION:
This study is planned to be a prospective observational clinical study. Patients who will undergo on-pump coronary artery bypass surgery, meet the eligibility criteria and agree to participate in the study and sign the informed patient consent form will be included in the study.Systemic immune inflammatory index, systemic inflammatory response index, neurophile lymphocyte ratio, platelet lymphocyte ratio will be calculated in the routine complete blood count of patients in the last 3 preoperative days and in the first 24 hours postoperatively.It will be evaluated whether these biomarkers are related to the anesthesia technique used, patients comorbidities and the complications that develop in the first 24 hours postoperatively. Patients will be evaluated preoperatively, intraoperatively and postoperatively; preoperative comorbidities, intraoperative anesthesia management, cross clamp, pump and surgery times, blood and blood product transfusion, inotrope use and complications that develop up to the first 24 hours postoperatively will be recorded.The anesthetic technique to be used will be determined according to the anesthesiologist's preference and will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* On-pump bypass surgery
* Del-Nido cardioplegia used in operation
* ASA (American Society of Anesthesiologists) II- III patients

Exclusion Criteria:

* Patients with active malignancy
* Diagnosed with systemic inflammatory disease or autoimmune disease
* Chronic liver and kidney disease
* History of cerebrovascular disease within 6 months
* EF (Ejection Fraction) < 45%
* Non-cooperative or patients who do not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA (American Society of Anesthesiologists) II- III patients over the age of 18 who will undergo on-pump bypass surgery in Ankara City Hospital Bilkent and who agree to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Preoperative systemic immune inflammatory index (SII) | within 3 days preoperatively
  It will be calculated as: platelet count x neutrophil count / lymphocyte count from routine complete blood count
Postoperative systemic immune inflammatory index (SII) | in the first 24 hours postoperatively
  It will be calculated as: platelet count x neutrophil count / lymphocyte count from routine complete blood count
Preoperative systemic inflammatory response index (SIRI) | within 3 days preoperatively
  It will be calculated as: neutrophil count x monocyte count/lymphocyte count from routine complete blood count
Postoperative systemic inflammatory response index (SIRI) | in the first 24 hours postoperatively
  It will be calculated as: neutrophil count x monocyte count/lymphocyte count from routine complete blood count
Preoperative neutrophile lymphocyte ratio (NLR) | within 3 days preoperatively
  It will be calculated as:neutrophil count/lymphocyte count from routine complete blood count
Postoperative neutrophile lymphocyte ratio (NLR) | in the first 24 hours postoperatively
  It will be calculated as:neutrophil count/lymphocyte count from routine complete blood count
Preoperative platelet lymphocyte ratio (PLR) | within 3 days preoperatively
  It will be calculated as: platelet count/lymphocyte count from routine complete blood count
Postoperative platelet lymphocyte ratio (PLR) | in the first 24 hours postoperatively
  It will be calculated as: platelet count/lymphocyte count from routine complete blood count
Preoperative c-reactive protein | within 3 days preoperatively
  from routine preoperative blood sample ( milligram/decilitre)
Preoperative procalcitonin | within 3 days preoperatively
  from routine preoperative blood sample ( microgram/litre)
Postoperative c-reactive protein | in the first 24 hours postoperatively
  from routine postoperative blood sample ( milligram/decilitre)
Postoperative procalcitonin | in the first 24 hours postoperatively
  from routine postoperative blood sample ( microgram/litre)
Postoperative complications | within the first 24 hours after surgery
  Postoperative complications consisting of:
  * newly developed atrial fibrillation
  * need for cardiac pacing
  * need for ECMO (Extracorporeal membrane oxygenation)
  * need for IABP (Intra-Aortic Balloon Pump)
  * prolonged mechanical ventilation
  * pericardial effusion
  * cardiac arrest
  * cerebrovascular event
  * delirium
  * exitus
  * other complications.

SECONDARY OUTCOMES:
Patient comorbidities | preoperative within 48 hours
  Patient comorbidities will be assessed
Transfusion requirement | during the operation
  Incidence of transfusion of blood and blood products to the patient
Inotrope requirement | during the operation
  Incidence of inotrope usage, inotropes consisting of:
  * noradrenaline
  * dopamine
  * dobutamine

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara city hospital bilkent, Ankara, Çankaya, Turkey (Türkiye)